CLINICAL TRIAL: NCT04152109
Title: Evaluation of Integrative and Complementary Practices in Health (PICS)
Brief Title: Integrative and Complementary Health Practices (PICS)
Acronym: PICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Triangulo Mineiro (Other)
Responsible Party: Principal Investigator, Elida Mara Carneiro da Silva, Doctor of Health Sciences, Universidade Federal do Triangulo Mineiro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Elida123
Record Dates: First submitted 2019-09-21; First posted 2019-11-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Neoplasms; Epilepsy
Keywords: complementary medicine; laying on of hands; cancer; epilepsy; complementary therapies
MeSH Terms: conditions — Neoplasms; Epilepsy | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigators and outcome evaluators will be blind to interventions that participants receive (do not know participants' allocation) and participants will be blind to subgroups without laying on of hands, laying on of hands with and without Spiritual connection (Spirit "passe"), not knowing which group they were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Without laying on of hands (Other): The patients will remain in bed supine with blindfolds. A volunteer will move close to the patient with hands behind and mentally repeat the alphabet or do count math during 5 minutes, around 8 weeks.
  Interventions: Other: Without laying on of hands subgroup
- Laying on of hands with healing intent and without Spiritual connection (Sham Comparator): Participants included in this subgroup will be exposed to the laying on of hands with healing intent by volunteers. The patients will be blindfold in the supine bed during 5 minutes, 8 weeks.
  Interventions: Other: Laying on of hands without Spiritual connection
- Laying on of hands with healing intent and Spiritual connection by Spiritual "Passe" (Experimental): The participants will be subjected application of the laying on of hands by the passistas who will give the Spiritist "passe". Patients remain in the supine bed blindfolded for 5 minutes, around 8 weeks.
  Interventions: Other: Laying on of hands by Spiritual "Passe"

INTERVENTIONS:
Other: Without laying on of hands subgroup — The patients will remain in bed supine with blindfolds. A volunteer will move close to the patient with hands behind and mentally repeat the alphabet or count during 5 minutes, around 8 weeks.
  Arms: Without laying on of hands
Other: Laying on of hands without Spiritual connection — Participants included in this subgroup will be exposed to the laying on of hands with healing intent by volunteers. The patients will be blindfold in the supine bed during 5 minutes, around 8 weeks.
  Arms: Laying on of hands with healing intent and without Spiritual connection
Other: Laying on of hands by Spiritual "Passe" — The participants will be subjected application of the laying on of hands by the volunteer who will give the Spiritist "passe". Patients remain in the supine bed blindfolded for 5 minutes, around 8 weeks.
  Arms: Laying on of hands with healing intent and Spiritual connection by Spiritual "Passe"

SUMMARY:
Complementary medicine, considered an unconventional approach, is performed in conjunction with conventional medicine. In Brazil, Integrative and Complementary Practices in Health have been inserted by the National Ordinance of Integrative and Complementary Practices. The aim of this study is to evaluate the effects of laying on of hands with spiritual connection by the Spiritist Passe about mental and physical health and quality of life of individuals.

DETAILED DESCRIPTION:
Type of study: randomized controlled trial. The sample will consist of cancer and epileptic patients including individuals aged eigtheen years and over. Patients will be referred by health professionals and social workers from Lar da Charidade, Clinics Hospital and attachments, as well as from the general community and will be invited to participate in the study at the Center for Integrative and Complementary Practices of the Clinics Hospital.

Participants will answer the questionnaires before the start of the study, after eight sessions and fiveteen days or the end of the research according to the group. The participants will be submitted to blood collection, when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients: diagnosis of neoplasia receiving parenteral chemotherapy.
* Epileptic patients: clinical diagnosis of focal epilepsy

Exclusion Criteria:

* Cancer patients: pregnant women, unable to understand the questionnaires; non-attendance of 3 sessions of therapy application and refusal to sign the consent form.
* Epileptic patients: people unable to understand the questionnaires; non-attendance of 3 sessions of therapy application and refusal to sign the consent form, as well as special groups (pregnant women, newly diagnosed epilepsy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2025-12-02 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Evaluation of Anxiety by Depression, Anxiety and Stress Scale. Scores between 0-63. Higher score indicates greater severity.
Stress | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Evaluation of stress by Depression, Anxiety and Stress Scale. Scores between 0-63. Higher score indicates greater severity.
Depression | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Evaluation of Depression by by Depression, Anxiety and Stress Scale. Scores between 0-63. Higher score indicates greater severity.

SECONDARY OUTCOMES:
Fatigue cancer patients | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Functional Assessment of Chronic Illness Scale. Higher score on the scale indicates greater fatigue level.
Quality of life in cancer patients | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Questionnaire developed to assess the quality of life of cancer patients. Lower score by scale indicates poorer quality of life.
Analysis of blood | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Blood collection for complete blood count.
Assessment of blood pressure | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Blood pressure, measured by the BPA 100 Microlife automatic oxygenation device
Assessment of peripheral oxygen saturation | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Peripheral oxygen saturation by the fingertip handheld pulse oximeter
Assessment of heart rate | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Heart rate (HR) by the fingertip handheld pulse oximeter.
Quality of life in epileptic patients | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Quality of life in epileptic patients by EQ-5D
Fatigue in epileptic and cancer patients | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Fatigue in epileptic and cancer patients by Fatigue pictogram. Scores between 0 - 4.
Brain electrical activity in epileptic patients | Change from Baseline the results anxiety at 8 weeks.
  Assessment of brain electrical activity in epileptic patients by electroencephalogram.
Pain intensity | Change from Baseline the results anxiety at 8 weeks and maintained at 10 weeks.
  Assessment of pain by Visual pain scale (VAS). Scores between 0 - 10. High scores indicates worse pain intensity.
Autonomic Response in epileptic patients | Change from Baseline the results anxiety at 8 weeks.
  Assessment of Heart rate variability by electrocardiogram with assessment of heart rate variability.

CONTACTS AND LOCATIONS:
Locations (1):
- Núcleo de Praticas Integrativas e Complementares, Uberaba, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No